CLINICAL TRIAL: NCT03425357
Title: Responsiveness of Sonoelastography in the Supraspinatus Tendon
Brief Title: Sonoelastography of the Supraspinatus Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Brage (Other)
Collaborators: Odense University Hospital (Other); Sygehus Lillebaelt (Other); Gigtforeningen (Other); Region of Southern Denmark (Other); Radiograf Rådet (Unknown)
Responsible Party: Sponsor-Investigator, Karen Brage, Ph.D-student, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sonoelastography_Supraspinatus
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Elasticity Imaging Techniques; Tendinopathy; Rotator Cuff Tendinitis; Musculoskeletal Disease
MeSH Terms: conditions — Tendinopathy; Rotator Cuff Injuries; Musculoskeletal Diseases | interventions — Exercise; Physical Therapy Modalities; Posture; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Load Exercises (Experimental): An exercise program consisting of 6 active exercises. Two exercises for the rotator cuff: Full Can and Sidelying external rotation Two exercises for the scapulae stabilizing muscles: Low Row and Push-Up Plus Two glenohumeral/postural corrective exercises: Posterior GH stretch and Scapular Retraction.
  Interventions: Other: Low Load Exercises

INTERVENTIONS:
Other: Low Load Exercises — All rotator cuff and scapular exercises are performed with 3 sets of 20 repetitions 3 times per week for 12 weeks. The load is set at around 60% of 1 RM (20 reps).
  The glenohumeral/postural corrective exercises are performed with 3 sets of 5 repetitions (The position is held for 15 seconds per repetition).
  Other Names: Scapular stabilization; Rotator Cuff; Exercise; Physiotherapy; Posture; Progressive exercise; Strength training

SUMMARY:
This study aims a determine the responsiveness of sonoelastography in the tendinopathy-affected supraspinatus tendon.

DETAILED DESCRIPTION:
The trial will include 20 patients diagnosed with supraspinatus tendinopathy from one orthopaedic shoulder clinic in Denmark.

The intervention will consist of an exercise program including lowload exercises with elastics and dumbbells, targeting the rotator cuff in a 12 weeks home-exercise program with two control visits at a physiotherapy department at the hospitals.

Tissue elasticity (measured by sonoelastography) is used as the primary outcome and is measured 12 weeks post baseline

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand Danish
* Shoulder pain > 3 months
* Positive on 3/5 clinical tests (full can, empty can, resisted external rotation, neers, hawking)
* Tendinopathy (MRI)

Exclusion Criteria:

* BMI > 30
* Bilateral shoulder pain
* Supraspinatus full thickness rupture (US)
* Biceps rupture (US)
* Calcification in supraspinatus (X-ray)
* Pregnancy
* Glenohumeral arthrosis (X-ray)
* Frozen shoulder
* Shoulder symptoms originating from neck
* Shoulder fracture, operation or luxation
* Known neuromuscular disease, rheumatoid arthritis, cancer, fibromyalgia, spondylarthropathy or psychiatric disorders
* Labrum lesion (MRI)
* Tear (˃1/3 of supraspinatus, vertical height) (MRI)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Tendon quality (SEL) | Baseline and 12 weeks
  Change from baseline in tendon quality (sonoelastography - strain elasticity)

SECONDARY OUTCOMES:
Tendon quality (MRI) | Baseline and 12 weeks
  Change from baseline in tendon quality (MRI)
Tendon quality (US) | Baseline and 12 weeks
  Change from baseline in tendon quality (conventional ultrasound)
Strength | Baseline and 12 weeks
  Change from baseline in Isometric Strength (MVC)
Recovery | 12 weeks
  Change from baseline in Global Perceived Effect (GPE). Ranging from -3 to +3; - being a worsening, 0 being no change and + being an improvement.
Pain | Baseline and 12 weeks
  Change from baseline in Visual Analogue Scale (VAS). Ranging from 0 to 10; 0 being no pain and 10 being severe pain.

OTHER OUTCOMES:
Quality of life | Baseline and 12 weeks
  Change in Euro Qol 5D index (EQ-5D-3L). The system consists of a descriptive system and a visual analogue scale (EQ VAS). The descriptive system contains 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 3 levels; no problems, some problems and extreme problems. The EQ-VAS range from 0 (worst imaginable health state) to 100 (best imaginable health state).
Disability | Baseline and 12 weeks
  Change in Disability of the Arm, Shoulder and Hand questionnaire (DASH). Each item is rated with a score from 1 (least disability) to 5 (most disability). All scores are added together, producing a raw score, which is then transformed into a score of 100 maximum. A higher score indicates greater disability.
Demographic | Baseline
  Gender, age, bmi, education (level), duration of symptoms, symptom history

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Juul-Kristensen, Assoc Prof, Study Director — Department of Sport Science and Biomechanics
Locations (1):
- University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Brage K, Juul-Kristensen B, Hjarbaek J, Boyle E, Kjaer P, Ingwersen KG. Strain Elastography and Tendon Response to an Exercise Program in Patients With Supraspinatus Tendinopathy: An Exploratory Study. Orthop J Sports Med. 2020 Dec 16;8(12):2325967120965185. doi: 10.1177/2325967120965185. eCollection 2020 Dec. PMID 33403207